CLINICAL TRIAL: NCT01972139
Title: Renal Denervation Using the SYMPLICITY Renal Denervation System in Patients With Uncontrolled Hypertension - SYMPLICITY HTN-4
Brief Title: Renal Denervation in Patients With Uncontrolled Hypertension - SYMPLICITY HTN-4
Acronym: HTN-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HTN-4
Record Dates: First submitted 2013-10-22; First posted 2013-10-30 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Uncontrolled hypertension; blood pressure; renal denervation; HTN-4; SYMPLICITY
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation (Experimental): Subjects are treated with the renal denervation procedure after randomization.
  Interventions: Device: Renal Denervation using the Symplicity Renal Denervation System; Device: Renal Angiography
- Control (Other): Subjects randomized prior to enrollment closure were treated with sham renal denervation (angiography only). Once enrollment was closed and the protocol revised, no control subjects crossed-over.
  Interventions: Other: Sham Renal Denervation; Device: Renal Angiography

INTERVENTIONS:
Device: Renal Denervation using the Symplicity Renal Denervation System — Subjects randomized to the renal denervation group underwent angiography and renal denervation.
  Arms: Renal Denervation
Other: Sham Renal Denervation — Prior to enrollment closure, subjects were treated with sham renal denervation. After enrollment closure, subjects previously enrolled were no longer eligible to cross-over.
  Arms: Control
Device: Renal Angiography — Subjects who met all criteria after the screening period did undergo a renal artery angiogram to evaluate renal artery anatomy. Only subjects with eligible renal artery anatomy were randomized.

SUMMARY:
An international, multi-center, prospective, blinded, randomized, controlled trial. The objective is to demonstrate that catheter-based renal denervation is an effective and safe treatment for uncontrolled hypertension.

DETAILED DESCRIPTION:
After the 6 month follow-up required testing has been completed, control group subjects would be unblinded to their randomization group and would have an option, at the discretion of the Investigator and with written concurrence of the medical monitor, to be treated with renal denervation procedure. However, after enrollment closure, subjects previously randomized were no longer allowed to cross-over.

ELIGIBILITY:
Inclusion Criteria:

* Individual is on maximally tolerated stable medication regimen including 3 or more anti-hypertensive medications of different classes, one of which must be a thiazide or thiazide-like diuretic
* Individual has office SBP greater than or equal to 140mmHg and less than 160mmHg
* Individual has ABPM average SBP greater than or equal to 135 mmHg

Exclusion Criteria:

* Individual lacks appropriate renal artery anatomy
* Individual has eGFR of less than 30
* Individual has Type I diabetes mellitus
* Individual has had one or more episodes of orthostatic hypotension
* Individual requires chronic oxygen other than nocturnal respiratory support for sleep apnea
* Individual has primary pulmonary hypertension
* Individual has other concomitant conditions that may adversely affect the patient or the study outcomes
* Individual is pregnant, nursing or planning to be pregnant
* Individual has had a previous organ transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Reaching BP Goal | 6 months post-randomization
Incidence of Major Adverse Events through 1 month post-procedure (Renal artery stenosis measured at 6 months) | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute; Michael Weber, MD, Principal Investigator — SUNY Downstate College of Medicine
Locations (3):
- United States (3):
  - Piedmont Hospital, Atlanta, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina